CLINICAL TRIAL: NCT00703807
Title: A Phase I Study of the Weekly Oral RAD001 in Combination With Oral Topotecan in Patients With Advanced or Recurrent Endometrial Cancers
Brief Title: Study of the Weekly Oral RAD001 in Combination With Oral Topotecan in Patients With Advanced or Recurrent Endometrial Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Maysa Abu-Khalaf, Principal Investigator, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0804003747
Record Dates: First submitted 2008-06-20; First posted 2008-06-24 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Topotecan; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Daily oral RAD001 for 21 days in combination with oral topotecan on days 1-5 of a 21 day cycle
  Interventions: Drug: Topotecan; Drug: RAD001

INTERVENTIONS:
Drug: Topotecan — Dose escalation, 5 dose levels, 1.5 mg/m2 - 2.3 mg/m2, PO day 1-5 every 21 days
  Other Names: Hycamtin
Drug: RAD001 — Dose level -1, 5 mg qod Dose level 1, 5 mg qod Dose level 2, 5 mg qd Dose level 3, 5 mg qd DOse level 4, 10 mg qd
  Other Names: Everolimus

SUMMARY:
Endometrial cancer is the most common malignancy of the female reproductive tract. The majority of patients with endometrial cancer are diagnosed at an early stage and cured with surgery with or without adjuvant radiotherapy. However, a significant number of patients present with metastatic disease outside of the pelvis or develop recurrent disease after primary therapy.

mTOR inhibitors have been shown to be promising agents in reducing tumor growth in vitro and in vivo, in several solid cancers. Inhibitors of mTOR are primarily cytostatic in cancer cells; combination therapy with cytotoxic chemotherapeutics and other biologic agents may prove to be the most advantageous use of these drugs. mTOR inhibition with a rapamycin analogue demonstrated in vitro antiproliferative activity on endometrial AN3 CA and HEC-1-A tumor cells, and this inhibition of proliferation was found to be concentration dependent. Topotecan is an active agent in the treatment of advanced and recurrent endometrial cancers.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically-confirmed advanced or recurrent endometrial cancer
* Patients must be refractory to standard therapy or for which no curative standard therapy exists, to be considered. Metastatic disease, if present, should not be progressing so as to require palliative treatment within 4 weeks of enrollment based on clinical assessment by the investigator.
* Development of new lesions or an increase in preexisting lesions on bone scintigraphy, CT, MRI or by physical examination. Patients in whom the sole criterion for progression is an increase in a biochemical marker, e.g., carcinoembryonic antigen (CEA), or an increase in symptoms, are not eligible.
* Age ≥ 18 years
* WHO performance status ≤ 2
* Adequate bone marrow function as shown by: ANC ≥ 1.5 x 109/L, Platelets ≥ 100 x 109/L, Hb >9 g/dL
* Adequate liver function as shown by:
* serum bilirubin ≤ 1.5 x ULN
* INR < 1.3 (or < 3 on anticoagulants)
* ALT and AST ≤ 2.5x ULN (≤ 5x ULN in patients with liver metastases)
* Adequate renal function: serum creatinine ≤ 1.5 x mg/dL
* Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
* Signed informed consent

Exclusion Criteria:

* Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of study drug (including chemotherapy, radiation therapy, antibody based therapy, etc.)
* Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study
* Prior treatment with any investigational drug within the preceding 4 weeks
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent, except corticosteroids with a daily dosage equivalent to prednisone ≤ 20 mg. However, patients receiving corticosteroids must have been on a stable dosage regimen for a minimum of 4 weeks prior to the first treatment with RAD001. Topical or inhaled corticosteroids are allowed.
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:
* Symptomatic congestive heart failure of New York heart Association Class III or IV
* unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
* severely impaired lung function
* uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN
* active (acute or chronic) or uncontrolled severe infections
* liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* A known history of HIV seropositivity
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Patients with an active, bleeding diathesis
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. If barrier contraceptives are being used, these must be continued throughout the trial by both sexes. Hormonal contraceptives are not acceptable as a sole method of contraception. (Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to administration of RAD001)
* Patients who have received prior treatment with an mTOR inhibitor (sirolimus, temsirolimus, everolimus).
* Patients with a known hypersensitivity to RAD001 (everolimus) or other rapamycins (sirolimus, temsirolimus) or to its excipients
* History of noncompliance to medical regimens
* Patients unwilling to or unable to comply with the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To determine the safety, dose-limiting toxicities,and maximum tolerated dose of daily oral RAD001 in combination with oral topotecan given on days 1-5 q 21 days in patients with advanced or recurrent endometrial cancers | Upon completion of study

SECONDARY OUTCOMES:
To determine if daily administration of RAD001 changes the pharmacokinetic profile of oral topotecan, and if oral topotecan changes the pharmacokinetic profile of oral RAD001. | Upon completion of study
To determine the anti-tumor effect of the combination using Response Evaluation Criteria in Solid Tumors (RECIST) | Upon completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Maysa Abu-Khalaf, M.D., Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States